CLINICAL TRIAL: NCT00773279
Title: A Multi-centre, Randomised, Open-label, Cross-over Study to Explore Effectiveness, Safety, and Preference of a New Disposable Pen PDS290 Versus FlexPen® in Subjects With Type 1 or Type 2 Diabetes
Brief Title: Efficacy, Safety and Preference Study of a Insulin Pen PDS290 vs. a Novo Nordisk Marketed Insulin Pen in Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDS290-1971
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDS290 --> FlexPen® (Experimental): Subjects will receive trial drug with PDS290 for 12 weeks (treatment sequence 1) followed by FlexPen® for 12 weeks (treatment sequence 2)
  Interventions: Device: FlexTouch®; Device: FlexPen®
- FlexPen® --> PDS290 (Experimental): Subjects will receive trial drug with FlexPen® for 12 weeks (treatment sequence 1) followed by PDS290 for 12 weeks (treatment sequence 2)
  Interventions: Device: FlexTouch®; Device: FlexPen®

INTERVENTIONS:
Device: FlexTouch® — All subjects to receive insulin detemir treatment (and if relevant insulin aspart) with either a insulin pen PDS290 (FlexTouch®) or a Novo Nordisk marketed insulin pen (FlexPen®) for 12 weeks. After 12 weeks, all subjects will continue their insulin treatment with the other injection device.
Device: FlexPen® — All subjects to receive insulin detemir treatment (and if relevant insulin aspart) with either a insulin pen PDS290 (FlexTouch®) or a Novo Nordisk marketed insulin pen (FlexPen®) for 12 weeks. After 12 weeks, all subjects will continue their insulin treatment with the other injection device.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this clinical trial is to assess and compare the effect on blood sugar control of insulin detemir and insulin aspart or insulin detemir alone administered by a insulin pen PDS290 (FlexTouch®) versus a Novo Nordisk marketed insulin pen (FlexPen®) in subjects with type 1 or type 2 diabetes mellitus. Furthermore, the subject's preference of the devices will be investigated by the use of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Subjects diagnosed with type 1 or type 2 diabetes. If type 2 diabetics, treatment with or without oral anti diabetic medication is allowed
* Current users of vial/syringe (pen naïve) treated with short-acting insulin (insulin aspart, glulisine or lispro) and once daily long-acting insulin (detemir or glargine) or once daily long-acting insulin (detemir or glargine) alone
* Treatment with insulin (i.e. aspart, glulisine, lispro, detemir or glargine) for at least 6 months
* Body Mass Index (BMI) less than 45.0 kg/m^2
* HbA1c less than or equal to 9.0% at screening visit based on analysis from central laboratory
* Able and willing to adhere to the trial-specific insulin regimen for the entire trial period

Exclusion Criteria:

* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or inadequate contraceptive techniques during the trial period (adequate contraceptive measures are considered as intrauterine device, oral contraceptives and barrier methods)
* Previous participation in this trial (screening visit)
* Systemic drugs that may influence glycaemic control (e.g., corticosteroids)
* Known or suspected allergy to trial product(s) or related products
* Known or suspected abuse of alcohol or drug abuse
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Previous treatment with sitagliptin
* Clinically significant, active (or over the past 12 months) disease of the gastrointestinal, neurological, genitourinary, or haematological systems
* Cardiac disease defined as: Decompensated heart failure (New York Heart class III or IV, unstable angina pectoris within the past 6 months of study enrolment, myocardial infarction within the past 12 months and a clinically significant history of arrhythmias or conduction delays on electrocardiogram (ECG) over the past 12 months
* Any other severe acute or chronic illness as judged by the Investigator
* Recurrent major hypoglycaemia (defined as severe central nervous system dysfunction associated with hypoglycaemia, requiring the assistance of another person) or hypoglycaemia unawareness (defined as a condition in which subjects no longer experience the usual warning signs of hypoglycaemia; the symptoms of hypoglycaemia may be different, less pronounced or even absent) or hospitalisation for diabetic ketoacidosis during the previous six months
* Any other conditions that the Investigator judges would interfere with trial participation or evaluation of results (i.e. planned any diagnostic or therapeutic medical intervention such as surgery)
* Participated in another clinical trial and received an investigational drug within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (62):
- United States (62):
  - Novo Nordisk Investigational Site, Burlingame, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Salinas, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Lafayette, Indiana
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Bowling Green, Kentucky
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Tabor City, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Gallipolis, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Carlisle, Pennsylvania
  - Novo Nordisk Investigational Site, Little River, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Wielandt JO, Niemeyer M, Hansen MR, Bucher D, Thomsen NB. An assessment of dose accuracy and injection force of a novel prefilled insulin pen: comparison with a widely used prefilled insulin pen. Expert Opin Drug Deliv. 2011 Oct;8(10):1271-6. doi: 10.1517/17425247.2011.615308. Epub 2011 Sep 2. PMID 21883036
- [Result] Garg S, Bailey T, DeLuzio T, Pollom D. Preference for a new prefilled insulin pen compared with the original pen. Curr Med Res Opin. 2011 Dec;27(12):2323-33. doi: 10.1185/03007995.2011.630721. Epub 2011 Oct 31. PMID 21988614
- [Result] Nadeau DA, Campos C, Niemeyer M, Bailey T. Healthcare professional and patient assessment of a new prefilled insulin pen versus two widely available prefilled insulin pens for ease of use, teaching and learning. Curr Med Res Opin. 2012 Jan;28(1):3-13. doi: 10.1185/03007995.2011.644427. Epub 2011 Dec 20. PMID 22114905
- [Result] Hemmingsen H, Niemeyer M, Hansen MR, Bucher D, Thomsen NB. A prefilled insulin pen with a novel injection mechanism and a lower injection force than other prefilled insulin pens. Diabetes Technol Ther. 2011 Dec;13(12):1207-11. doi: 10.1089/dia.2011.0110. Epub 2011 Aug 24. PMID 21864019
- [Result] Bailey T, Thurman J, Niemeyer M, Schmeisl G. Usability and preference evaluation of a prefilled insulin pen with a novel injection mechanism by people with diabetes and healthcare professionals. Curr Med Res Opin. 2011 Oct;27(10):2043-52. doi: 10.1185/03007995.2011.616190. Epub 2011 Sep 14. PMID 21916529
- [Result] Oyer D, Narendran P, Qvist M, Niemeyer M, Nadeau DA. Ease of use and preference of a new versus widely available prefilled insulin pen assessed by people with diabetes, physicians and nurses. Expert Opin Drug Deliv. 2011 Oct;8(10):1259-69. doi: 10.1517/17425247.2011.615830. Epub 2011 Sep 12. PMID 21905942
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 61 sites in the United States of America (USA).
Pre-assignment Details: Screening period of 2 weeks where the subjects were assessed for eligibility, run-in period of 6 weeks, hereafter eligible subjects were randomised to one of the two 12-week treatment sequences: PDS290 -> FlexPen® or FlexPen® -> PDS290.
Period: Period 1
Arm/Group | PDS290 -> FlexPen® | FlexPen® -> PDS290
Started | 121 | 121
Completed | 114 | 117
Not Completed | 7 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Unclassified | 5 | 1
Period: Period 2
Arm/Group | PDS290 -> FlexPen® | FlexPen® -> PDS290
Started | 114 | 117
Completed | 111 | 111
Not Completed | 3 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 3
Not completed — Unclassified | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Entire Trial Population: Participants who in random order received usual insulin treatment with pre-filled pen device PDS290 for 12 weeks followed by switch to pre-filled pen device FlexPen® for 12 weeks or vice versa. The frequency of basal and bolus injections were kept the same throughout the trial. Both prefilled pens were self-administered subcutaneously by the participants.
Arm/Group | Entire Trial Population
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 226
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 199
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 242
HbA1c (glycosylated haemoglobin) [Mean (Standard Deviation); unit: percentage (%) of total haemoglobin] | 7.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin) for Participants Treated With PDS290 and FlexPen®
Time Frame: Week 12 of each treatment sequence
Population: Intention-to-treat (ITT) population comprising all randomised subjects and with data on HbA1c. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®). Some subjects dropped out during either treatment sequence.
Measure: Mean (Standard Deviation); unit: percentage (%) of total haemoglobin
Groups:
- PDS290: Participants who received usual insulin treatment with pre-filled pen device PDS290 (FlexTouch®).
- FlexPen®: Participants who received usual insulin treatment with pre-filled pen device FlexPen®.
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 232 | 233
percentage (%) of total haemoglobin | 7.5 (1.0) | 7.5 (1.0)
Statistical Analysis 1: Comparison: PDS290 vs FlexPen®; The null hypothesis is that PDS290 be not non-inferior to FlexPen® with respect to HbA1c after 12 weeks of treatment; non-inferiority margin is 0.4 % (absolute); Test type: Non-Inferiority or Equivalence — A two-sided 95 % Confidence Interval (CI) for the treatment difference, "PDS290 minus FlexPen", in HbA1c after 12 weeks of treatment. PDS290 was to be declared non-inferior to FlexPen® if the upper limit of that CI would be less than the non-inferiority margin 0.40 % (absolute); Linear mixed effect model; Linear mixed effect model with period and delivery systems as fixed effects, and subject as a random effect; Mean Difference (Final Values) = -0.047, 95% CI [-0.127 to 0.032], Standard Error of Mean 0.040

2. Secondary Outcome: Percentage of Subject Having Preference for PDS290 Versus FlexPen® in Terms of Convenience and Ease of Use
Description: Questionnaire (Niskanen Comparative Device Questionnaire) compared preference / convenience and ease of use by device specific questionnaire (summarised by scores of question 9)
Time Frame: Week 24
Population: ITT population. Some subjects did not have any available Niskanen Comparative Device Questionnaire results.
Measure: Number; unit: percentage of participants
Arm/Group | Entire Trial Population
Number analyzed (Participants) | 227
percentage of participants
  Preference of PDS290 | 68
  Preference of FlexPen® | 19
  No preference | 13

3. Secondary Outcome: Summary Score for Treatment Satisfaction
Description: Overall summary from Insulin Treatment Satisfaction Questionnaire (ITSQ) with higher scores (0-100) indicating greater satisfaction.
Time Frame: Week 24
Population: ITT population. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®). Some subjects did not have any available ITSQ results in PDS290 and FlexPen® treatment groups, respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 222 | 223
scores on a scale | 80.9 (11.3) | 76.8 (15.2)

4. Secondary Outcome: Score for Treatment Impact Measure for Diabetes
Description: Treatment Related Impact Measure for Diabetes (TRIM-D and TRIM-D device) with scores from 0-100, higher scores indicate less treatment related impact.
Time Frame: Week 24
Population: ITT population. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®). Some subjects did not have any TRIM-D available results in PDS290 and FlexPen® treatment groups, respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 232 | 232
scores on a scale
  TRIM-D total scores | 75.1 (13.1) | 72.8 (13.6)
  TRIM-D device scores | 84.9 (12.7) | 78.6 (16.6)

5. Secondary Outcome: Clinical Technical Complaints (CTCs)
Description: A clinical technical complaint is any written, electronic or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety or performance of a medical device.
Time Frame: Weeks 0-24 (whole trial period)
Population: ITT population. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®). Some subjects did not have any available results in PDS290 and FlexPen® treatment groups, respectively.
Measure: Number; unit: CTCs
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 242 | 242
CTCs | 67 | 84

6. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Presented by severity: major: subject not able to treat himself; minor: plasma glucose below 3.1 mmol/L; symptoms only: no plasma glucose measured or above or equal to 3.1 mmol/L.
Time Frame: Weeks 0-12 (first treatment) and 12-24 (second treatment)
Population: as for outcome 5
Measure: Number; unit: episodes
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 239 | 235
episodes
  All episodes | 1108 | 1092
  Major episodes | 7 | 3
  Minor episodes | 920 | 927
  Symptoms only | 181 | 162

7. Secondary Outcome: Number of Adverse Device Effects
Description: Adverse device effects were defined as clinical technical complaints (CTCs) related to an Adverse Event/Serious Adverse Event. This was defined as an adverse unintended reaction to a medical device. This definition includes any event which is caused by an inadequate or incomplete user instruction or guide in the use of the device and any event caused by wrongful use.
Time Frame: From randomisation (week 0) and until 7 days after Week 24 (Visit 16)
Population: as for outcome 5
Measure: Number; unit: events
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 239 | 235
events | 0 | 0

8. Secondary Outcome: Hypoglycaemic Episodes, Number of Events Per Subject Day
Time Frame: Weeks 0-12 (first treatment) and 12-24 (second treatment)
Population: ITT population. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®).
Measure: Number; unit: events per subject-day
Arm/Group | PDS290 | FlexPen®
Number analyzed (Participants) | 239 | 235
events per subject-day | 0.06 | 0.06

ADVERSE EVENTS:
Time Frame: From randomisation and until seven days after Week 24 (Visit 16).
Description: ITT population. This was a cross-over trial, so subjects received treatment with both PDS290 and FlexPen®. Results are reported separately for each treatment period, i.e. PDS290 versus FlexPen®).
Arm/Group | PDS290 | FlexPen®
Serious Adverse Events (participants affected / at risk) | 7/238 | 5/235
Other Adverse Events (participants affected / at risk) | 25/238 | 31/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDS290 (N=238) | FlexPen® (N=235)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDS290 (N=238) | FlexPen® (N=235)
Nasopharyngitis (Infections and infestations) | 15 (19) | 20 (24)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (12) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data until specified milestones, eg a clinical trial report is available. This includes the right not to release interim results from clinical trials, because such results may lead to conclusions that are later shown to be incorrect. Novo Nordisk will not suppress or veto publications; however Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.